CLINICAL TRIAL: NCT01157468
Title: Study of Catalytic Antibodies in a Cohort Population of Martinique
Brief Title: Catalytic Antibodies and Lupus in Martinique
Acronym: LUMAB2
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 10/E/12
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus in Martinique; Hydrolase and DNase activities
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * For the "case" means the research will be done on a blood sample of 7 ml, reclassified from treatement to research, collected from the blood sampling usually prescribed by doctors to treat the patient come to be diagnosed a lupus or for continuing care.
  * For the "control" means research will be done on a blood sample of 7 ml collected from people coming to donate blood at thethe French Blood Establishment of Martinique.
  The volume does not exceed the maximum amount allowed by French regulations for blood donation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: The "Case" group is constituted with patients with Systemic Lupus Erythematosus from Martinique, divided en 2:
  * 30 patients with a quiescent lupus
  * 30 patients with an active lupus
- Controles: The "Control" group is constituted by people coming to give blood to the French Blood Establishment of Martinique.

SUMMARY:
* The Martinique island (French West-Indies) is an area of high prevalence and incidence for Systemic Lupus Erythematosus (SLE), respectively 64,2/ 100000 and 4,7/ 100000. In many cases, this disease concerns Afro Caribbean women, whose auto-antibodies are excessively high; also, organic damages are frequent. The disease can be fatal.
* Studies have shown that some cytotoxic auto-antibodies may have a responsibility in the hydrolysing of DNA. This study will focus on the DNA activity and also on the overwhelm hydrolase activity dealing with the Lupus disease in order to measure the link between the disease activity and the catalytic activity. Patients concerned by this study will be Martinique people.

DETAILED DESCRIPTION:
This study will be conducted as an case-control survey.

* The first group with patients: 60 SLE patients, 30 patients with a quiescent lupus and 30 patients with an active lupus. Patients that will be included are followed by the University hospital of Fort-de-France.
* The second group is the control group: subjects will be recruited by the French organisation responsible for donation of blood.

Test will be done at the UMRS 872 laboratory of the INSERM - Laboratory of Immunopathology and Therapeutic immunointervention - in Paris ; two catalytic activities will be tested: the DNase activity and the hydrolase activity.

Means to analyse the two activities: digestion of plasmid and Affinity-linked Oligonucleotide Nuclease Assay for DNase activity and hydrolysis of a peptide PFR-MCA for hydrolase activity.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Presence of systemic lupus erythematosus according to the criteria of the modified 1997 ARA 1982 Lupus systemic evolution: Rates of anti DNA> 100 U/L in ELISA and SLEDAI> 7. Quiescent systemic Lupus: SLEDAI <7
* Be aged 18 years and over
* Patient who has his main home in Martinique
* Patient who gave his agreement to participate in this clinical study

For control subjects:

* Voluntary donor who gave freely his agreement to participate in this study
* Be aged 18 years and over
* Patient who has his main home in Martinique
* Voluntary who gave his agreement to participate in this clinical study

Exclusion Criteria:

For patients:

* Presence of mixed connective tissue disease, Hashimoto
* Patients with other diseases: cancer, current infection
* Patient pregnant or breast-feeding
* Patient who refuse to participate in the study
* Patient not affiliated with a social security scheme (beneficiary or beneficiary)
* Specially Protected Persons (or under guardianship)
* Patient who has not his main home in Martinique

For control subjects:

* Voluntary donor who refused to participate in this study
* Voluntary who has not main home in Martinique

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases are patients with Systemic Lupus Erythematosus treated at the Centre Hospitalier of Fort de France (Martinique): patients with a quiescent lupus and patients with an active lupus.
  Controles are people coming to donate blood samples at the French Blood Establishment of Martinique.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency of hydrolase and DNase activities | 2 years
  Estimate the presence of a significant enzymatic activity by calculating the frequency of the hydrolase and DNase activities in lupus in Martinique(French west-indies)

SECONDARY OUTCOMES:
Association of disease activity and catalytic activity | 2 years
  Evaluate the strength of the association of disease activity and catalytic activity of antibodies (quiescent / active and control / patient)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DELIGNY, MD, Principal Investigator — Service de Médecine Interne - Centre Hospitalier Universiatire de Fort de France
Locations (1):
- Centre Hospitalier Universitaire de Fort de France, Fort de France, Martinique, France